CLINICAL TRIAL: NCT01492933
Title: Measuring Effects of Acute Ethanol on Human Brain Metabolites Using Magnetic Resonance Spectroscopy
Brief Title: Measuring Effects of Alcohol on Brain Chemistry
Status: Terminated | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120032; 12-AA-0032
Record Dates: First submitted 2011-12-14; First posted 2011-12-15 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2015-02-24

CONDITIONS: Healthy Volunteers
Keywords: Ethanol; Magnetic Resonance Spectroscopy; Spectroscopy; Alcohol Use
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Studies show that alcohol changes the amount of many brain chemicals. These changes may be related to continued drinking, craving for alcohol, and relapse. This study will use magnetic resonance imaging (MRI) to look at brain areas and brain chemistry during an infusion of alcohol. It will also study how changes in brain chemistry relate to participant reports of feeling drunk.

Objectives:

- To use magnetic resonance imaging to measure the effect of alcohol on brain chemistry

Eligibility:

* Individuals between 21 and 45 years of age.
* Participants will be either light drinkers (1 to 14 standard alcoholic drinks per week) or heavy drinkers (20 to 40 standard alcoholic drinks per week). A standard drink is a 12-ounce beer, a 4-ounce glass of wine, or a shot of liquor.
* Participants must be able to go without alcohol for at least 3 days in a row without severe withdrawal symptoms.

Design:

* This study requires two or three outpatient visits to the NIH Clinical Center.
* Participants will have a physical exam and medical history. Blood and urine samples will be collected. Participants' alcohol drinking habits will also be assessed to determine whether they may have an alcohol use disorder.
* At the first study visit, participants will have an infusion of alcohol. Blood samples will be collected to measure blood alcohol levels.
* The MRI study visit will take place about 3 days after the first study visit. Participants will have an MRI scan of the brain, followed by an infusion of alcohol and another scan. Blood samples will be collected.
* Participants will complete questionnaires before and after each infusion to measure their response to alcohol.
* Heavy drinkers will come to the clinic for a third visit to discuss possible future treatment and any risky behavior associated with their high levels of alcohol use.

DETAILED DESCRIPTION:
Rodent studies have indicated that modulation of glutamatergic transmission contributes to alcohol intoxication, reinforcement, tolerance, and dependence. Brain microdialysis studies have in general shown that acute alcohol suppresses glutamate release, while alcohol withdrawal leads to progressively increased extracellular levels.

Here, we will use an acute, pharmacokinetically controlled alcohol challenge and magnetic resonance spectroscopy (MRS) to study the relationship between brain alcohol and glutamate concentrations, and correlate these with subjective feelings of alcohol effects, as measured by the Drug Effects Questionnaire (DEQ) in human subjects. Correlations between MRS data and other behavioral data from the Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ), Alcohol Sensitivity Questionnaire (ASQ), and the Alcohol Effects Questionnaire (AEFQ) will be investigated.

Healthy participants aged 21-45, without gross impairment of judgment or complicated psychiatric or other morbidity, will receive a preliminary infusion to ensure no adverse effects from intravenous (IV) alcohol administration to a target BAC of 0.08g/dl. In a subsequent session, participants will be infused with alcohol to the same target level while being scanned in the MR scanner and reporting subjective feelings using the DEQ. Two groups of subjects will be recruited: heavy drinkers, classified as females who consume 15 plus drinks per week and males who consume 20 plus drinks per weekthose who consume between 20 and 40 drinks per week, and light drinkers, classified as females who consume between 1 and 10 drinks per week and males who consume between 1 and 14 drinks per week. those who consume between 1 and 14 drinks per week.

Central glutamate levels will be quantified at 3T using pharmacologically validated MRS methodology recently published from our laboratory, and its relationship to central alcohol levels will be determined. Relationships will also be analyzed between DEQ scores and brain glutamate and alcohol levels. Finally, it will be examined whether drinking history (i.e. being a light versus heavy drinker) is a moderator of any of these relationships.

ELIGIBILITY:
* INCLUSION CRITERIA (Light Drinkers)

  1. In good health as determined by medical history, physical exam, ECG and lab tests;
  2. Between 21 and 45 years of age;
  3. Currently consuming between 1 and 10 drinks per week for females and 1 and 14 drinks per week for males.

EXCLUSION CRITERIA (Light Drinkers)

1. Have liver function tests (AST, ALT, GGT, ALP) 3-times the upper limit of normal (ULN); or have Total Bilirubin above 1.5 ULN and Albumin below 3.5 g/dL.
2. Have fulfilled DSM-IV criteria for a current or past major psychiatric disorder including alcohol or other substance dependnece (excluding nicotine);
3. Have a Body Mass Index (BMI) value over 35;
4. Unable to stop taking any prescribed, non-prescribed, or over-the-counter medication or drugs 3 days prior to study days (excluding oral contraceptive agents). If a subject is taking a prescribed medication (excluding oral contraceptive agents) that is not take-as-needed they will be excluded from participation;
5. Are pregnant, as determined by a negative pregnancy test, or lactating;
6. Report to have a "facial flushing" response to the consumption of alcohol;
7. Have never consumed at least two standard drinks of alcohol within one hour;
8. Have ferromagnetic objects in their bodies, which might be adversely affected by MRI including implanted pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metal fragments in the eye that welders and other metal works may have any doubt about presence of these objects will result in exclusion from this study);
9. Regular tobacco users will be excluded from the study in order to avoid nicotine withdrawal symptoms. Occasional (not daily) use of tobacco products is acceptable;
10. Unwilling to abstain from alcohol for at least 2 days prior to the studies.

INCLUSION CRITERIA (Heavy Drinkers)

1. In good health as determined by medical history, physical exam, ECG and lab tests;
2. Between 21 and 45 years of age;
3. Currently consuming 15+ drinks for females and 20+ drinks for males;
4. Not regularly abstinent for more than 3 days per week, but have abstained from alcohol for 3 consecutive days without experiencing withdrawal symptoms;
5. Able to provide a plausible history that they can abstain from alcohol without significant withdrawal symptoms when coming to the clinic. In addition, participants will be asked to quantify their worst withdrawal symptoms using the Clinical Institute Withdrawal Assessment (CIWA) Instrument. Participants who score 8 or above will not be enrolled in the protocol;
6. Not seeking treatment for their alcohol consumption.

EXCLUSION CRITERIA (Heavy Drinkers)

1. Have liver function tests (AST, ALT, GGT, ALP) 3-times the upper limit of normal (ULN); or have Total Bilirubin above 1.5 ULN and Albumin below 3.5 g/dL.
2. Have fulfilled DSM-IV criteria for a current or past major psychiatric disorder, including any substance dependence (excluding alcohol or nicotine) at any time;
3. Have a Body Mass Index (BMI) value over 35;
4. Unable to stop taking any prescribed, non-prescribed, or over-the-counter medication or drugs 3 days prior to study days (excluding oral contraceptive agents). If a subject is taking a prescribed medication (excluding oral contraceptive agents) that is not take-as-needed they will be excluded from participation;
5. Are pregnant, as determined by a negative pregnancy test, or lactating;
6. Report to have a "facial flushing" response to the consumption of alcohol;
7. Have never consumed at least two standard drinks of alcohol within one hour;
8. Have ferromagnetic objects in their bodies, which might be adversely affected by MRI including implanted pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metal fragments in the eye that welders and other metal works may have any doubt about presence of these objects will result in exclusion from this study);
9. Regular tobacco users will be excluded from the study in order to avoid nicotine withdrawal symptoms. Occasional (not daily) use of tobacco products is acceptable;
10. Unwilling to abstain from alcohol for at least 2 days prior to the studies.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-11-22; Study Completion 2015-02-24

PRIMARY OUTCOMES:
What is the correlation between measured blood and breath alcohol level and ethanol level concentration computed from MRS. | End of study

SECONDARY OUTCOMES:
Does ethanol administration similarly affect the metabolite activities in all the regions of the brain Gray and White matter? | End of study
Measure: Does ethanol metabolite concentration correlate with any of subjective effects of ethanol as measured by response to DEQ questions? | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Reza Momenan, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Beckmann CF, Smith SM. Tensorial extensions of independent component analysis for multisubject FMRI analysis. Neuroimage. 2005 Mar;25(1):294-311. doi: 10.1016/j.neuroimage.2004.10.043. Epub 2005 Jan 8. PMID 15734364
- [Background] Romanos GE, Schroter-Kermani C, Bernimoulin JP. [Collagen as a basic element of the periodontium: immunohistochemical aspects in the human and animals. 2. Cementum and periodontal ligament]. Parodontol. 1991 Feb;2(1):47-59. German. PMID 1854918
- [Background] Behrens TE, Berg HJ, Jbabdi S, Rushworth MF, Woolrich MW. Probabilistic diffusion tractography with multiple fibre orientations: What can we gain? Neuroimage. 2007 Jan 1;34(1):144-55. doi: 10.1016/j.neuroimage.2006.09.018. Epub 2006 Oct 27. PMID 17070705